CLINICAL TRIAL: NCT02982980
Title: Muscle Strength Exercises After Breast Cancer Surgery: a Randomized Clinical Trial
Brief Title: Upper Limb Muscular Strengthening in the Rehabilitation of Patients Submitted to the Breast Cancer Surgical Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Gil Facina, Doctor, Federal University of São Paulo
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: FUSaoPauloPT5
Record Dates: First submitted 2016-12-02; First posted 2016-12-06 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-12

CONDITIONS: Muscle Strength Quantitative Trait Locus 1

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Physiotherapy Guidance Mastectomy (Experimental): Patients who underwent radical breast surgery, received pre and postoperative assessment and orientation.
  Interventions: Procedure: Physiotherapy Guidance
- Phys Muscle strengthening Mastectomy (Experimental): Patients who underwent radical breast surgery, in addition to receiving guidance, had, weekly, physical therapy sessions with the goal to increase muscle strength in the upper limbs, between one and three months after surgery.
  Interventions: Procedure: Physiotherapy Muscle strengthening
- Physiotherapy Guidance Quadrantectomy (Experimental): Patients who underwent partial breast surgery, received pre and postoperative assessment and orientation.
  Interventions: Procedure: Physiotherapy Guidance
- Phys Muscle strengthening Quadrantectomy (Experimental): Patients who underwent partial breast surgery, in addition to receiving guidance, had, weekly, physical therapy sessions with the goal to increase muscle strength in the upper limbs, between one and three months after surgery.
  Interventions: Procedure: Physiotherapy Muscle strengthening

INTERVENTIONS:
Procedure: Physiotherapy Guidance — Pre and postoperative assessment and orientation, guidelines for lymphedema prevention and self drainage, follow-up for rehabilitation or maintenance of joint amplitude of shoulder movements and functional return.
  Arms: Physiotherapy Guidance Mastectomy; Physiotherapy Guidance Quadrantectomy
Procedure: Physiotherapy Muscle strengthening — The exercises performed were active-free, with the aid of a stick or resistance by elastic bands and dumbbells for flexion, extension, adduction, abduction, external and internal rotation of the shoulder, and elbow flexion and extension, besides activities to enable movements Functional. The mode of execution of the exercises was isotonic, done slowly and within the joint amplitude reached by the patient, using resistance according to the muscular capacity of each patient.
  Arms: Phys Muscle strengthening Mastectomy; Phys Muscle strengthening Quadrantectomy

SUMMARY:
The presence of pain, reduced range of motion and decrease of muscle strength of the upper limb in the early postoperative period are some of the major deficiencies of the breast cancer patients.

The objectives of this study were to evaluate muscle strength, range of motion (ROM), pain, perimetry of the upper limbs and applied questionnaires of the upper lim function and quality of life, in patients after surgical treatment of breast cancer in different postoperative periods and different groups following rehabilitation: traditional postoperatively exercise to perform at home versus traditional exercises associated with weekly physiotherapy sessions to strength training for shoulder movements.

DETAILED DESCRIPTION:
A clinical trial, randomized, blinded study. The groups were divided according to the type of rehabilitation (weekly sessions of Physiotherapy-F and Orientation -O). The surgical type (M-Mastectomy and Q-Quadrantectomy) was also taken into account.

Were not included in the study those patients who underwent previous surgeries of breast cancer, breast reconstruction, those with some neurological deficit or acute orthopedic shoulder injury, such as tendonitis or bursitis, patients with previous histories of shoulder fracture with limited range of motion and tumor stage T4b or N3 or patients with bone or brain metastases.

All patients underwent preoperative evaluation and guidance of general care; then returned after one, two, three and six months postoperatively for reassessment and reorientation. The physiotherapy group, in addition to receiving guidance, had, weekly, physical therapy sessions with the goal to increase muscle strength in the upper limbs, between one and three months after surgery.The exercises performed were active-free, with the aid of a stick or resistance by elastic bands and dumbbells for flexion, extension, adduction, abduction, external and internal rotation of the shoulder, and elbow flexion and extension, besides activities to enable movements functional. The mode of execution of the exercises was isotonic, done slowly and within the joint amplitude reached by the patient, using resistance according to the muscular capacity of each patient.

All evaluations were performed by the physiotherapy team; the professionals were not aware of whether the patient belonged to the physiotherapy group or to the guidance group, constituted by a single evaluator (blinded study).

The evaluations were: muscular strength of the shoulder, evaluated by means of a manual isokinetic dynamometer, which records the peak of force, in kilograms, during five seconds of muscle contraction duration; range of motion of the shoulder: measured by a goniometer; function of the upper limb: ascertained by the application of a specific questionnaire, the Disabilities of the Arm, Shoulder and Hand Questionnaire (DASH) assesses functional capacity in upper limb diseases and measures the abilities to perform certain activities; pain: evaluated by the application of the Verbal Numerical Pain Scale (NVA); perimetry: evaluated with a tape measure in eight distinct points in the upper limbs and quality of life, analyzed by a European Organization for Research and Treatment of Cancer (EORTC) Quality of Life C30 (QLQ-C30) questionnaire with a Specific module for breast cancer (BR) 23 - Breast Specific Module.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing radical or conservative surgical treatment of breast cancer
* Patients who did some type of investigation of axillary lymph node involvement, sentinel lymph node biopsy (BLS) or lymph node dissection (LND)
* Patients who have performed the final and final evaluation
* Patients in the Muscular Strength group, who have not missed more than 3 treatment sessions

Exclusion Criteria:

* patients submitted to a new breast surgical intervention during the total time of follow-up of the research.
* previous surgeries of breast cancer;
* bilateral surgeries
* immediate breast reconstruction
* neurological deficit or acute orthopedic affection in the shoulder,
* advanced tumor stage T4b or N3 or patients with bone or brain metastases

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2011-08; Primary Completion 2012-08 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Muscle strength | two years
  Muscle strength of shoulder movements with Hand Held Dynamometer model 01163, Lafayette Instrument Company.

SECONDARY OUTCOMES:
Range of motion | two years
  Shoulder range of motion measured by a goniometer
Upper limb function | two years
  Upper limb function determined by the application of a specific questionnaire, the DASH (Disability of Arms, Shoulder and Hand Questionnaire)
Pain | two years
  Pain: assessed by the application of the Verbal Numerical Pain Scale (VN)
Perimeter | two years
  Perimeter: evaluated with a tape measure at eight distinct points in the upper limbs
Quality of life | two years
  Quality of life, analyzed by a questionnaire C30 (QLQ-C30) from the European Organization for Research and Treatment of Cancer (EORTC) Cancer, BR-23 (Breast Specific Module ).

CONTACTS AND LOCATIONS:
Overall Officials: Gil Facina, PhD, Principal Investigator — Federal University of São Paulo